CLINICAL TRIAL: NCT07005154
Title: A Phase 2, Open-label, Multi-cohort Study to Assess the Efficacy and Safety of ASP5541 in Participants With Advanced Prostate Cancer
Brief Title: A Phase 2 Study to Evaluate the Effects of ASP5541 in Participants With Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5541-CL-0201
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Metastatic Castration-Resistant Prostate Cancer; Metastatic Hormone Sensitive Prostate Cancer
Keywords: ASP5541; PRL-02
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone; Prednisolone; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (mCRPC) Group A (Experimental): Participants will receive ASP5541 every 12 weeks + prednisone/prednisolone twice daily
  Interventions: Drug: ASP5541; Drug: Prednisone; Drug: Prednisolone
- Cohort 1 (mCRPC) Group B (Active Comparator): Participants will receive abiraterone acetate once daily + prednisone/prednisolone twice daily
  Interventions: Drug: Prednisone; Drug: Prednisolone; Drug: abiraterone acetate
- Cohort 2 (mHSPC) Group A (Safety Run In) (Experimental): Participants will receive ASP5541 every 12 weeks
  Interventions: Drug: ASP5541
- Cohort 2 (mHSPC) Group B (Experimental): Participants will receive ASP5541 every 12 weeks
  Interventions: Drug: ASP5541
- Cohort 2 (mHSPC) Group C (Active Comparator): Participants will receive abiraterone acetate once daily + prednisone/prednisolone once daily
  Interventions: Drug: Prednisone; Drug: Prednisolone; Drug: abiraterone acetate
- Cohort 3 (mCRPC or mHSPC) Japanese Participants Only (Experimental): Participants will receive ASP5541 every 12 weeks + prednisone/prednisolone twice daily (for mCRPC) or prednisone/prednisolone once daily (for mHSPC)
  Interventions: Drug: ASP5541; Drug: Prednisone; Drug: Prednisolone

INTERVENTIONS:
Drug: ASP5541 — Intramuscular Injection
  Other Names: PRL-02
  Arms: Cohort 1 (mCRPC) Group A; Cohort 2 (mHSPC) Group A (Safety Run In); Cohort 2 (mHSPC) Group B; Cohort 3 (mCRPC or mHSPC) Japanese Participants Only
Drug: Prednisone — Oral
  Arms: Cohort 1 (mCRPC) Group A; Cohort 1 (mCRPC) Group B; Cohort 2 (mHSPC) Group C; Cohort 3 (mCRPC or mHSPC) Japanese Participants Only
Drug: Prednisolone — Oral
  Arms: Cohort 1 (mCRPC) Group A; Cohort 1 (mCRPC) Group B; Cohort 2 (mHSPC) Group C; Cohort 3 (mCRPC or mHSPC) Japanese Participants Only
Drug: abiraterone acetate — Oral
  Arms: Cohort 1 (mCRPC) Group B; Cohort 2 (mHSPC) Group C

SUMMARY:
Hormone therapy, or androgen deprivation therapy (ADT) is a standard way to treat prostate cancer. It works by reducing the amount of the main male sex hormone, testosterone in the body. Androgen receptor pathway inhibitors (ARPIs) are another type of hormone therapy. They either slow down how much testosterone is made or block testosterone from reaching the prostate cancer cells. Abiraterone acetate (AA) is an ARPI that is used to treat advanced prostate cancer. This type of treatment is usually given as a tablet with a steroid called prednisone/prednisolone to manage any medical problems from the hormone therapy. ASP5541 is a different form of AA. It is given as an injection into the muscle. In this study, ASP5541 will be given to men with advanced prostate cancer, both with and without prednisone/prednisolone. This study will check the safety of ASP5541 and compare how well ASP5541 works in men with advanced prostate cancer compared to AA.

The main aims of the study are to check how well ASP5541 with prednisone/prednisolone works compared to AA with prednisone/prednisolone in men with advanced prostate cancer who haven't previously been treated with an ARPI, to check safety of ASP5541 given by itself in men with advanced prostate cancer that haven't previously been treated with an ARPI, to check how well ASP5541 given by itself works compared to AA with prednisone/prednisolone in men with advanced prostate cancer that haven't previously been treated with an ARPI, and to check safety of ASP5541 with prednisone/prednisolone in Japanese men with advanced prostate cancer.

Adult men with a certain type of advanced prostate cancer can take part. Their cancer has spread to other parts of the body (metastatic). The different types are: Metastatic hormone-sensitive prostate cancer (mHSPC). Prostate cancer that needs testosterone to grow. Metastatic castration-resistant prostate cancer (mCRPC). Prostate cancer that continues to grow even when testosterone levels are low.

In this study there will be 3 treatment groups. In Group 1 men with mCRPC who haven't previously been treated with an ARPI will either be given ASP5541 and prednisone/prednisolone or AA and prednisone/prednisolone. In Group 2 men with mHSPC who haven't previously been treated with an ARPI will either be given ASP5541 by itself or be given AA with prednisone/prednisolone. In Group 3 Japanese men with mCRPC or mHSPC who may or may not have previously been treated with an ARPI will be given ASP5541 with prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Participant is diagnosed with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features.
* Participant has ECOG performance status of 0 or 1, or ECOG performance status of 2 if due to bone pain.
* Participant with mHSPC must have an estimated life expectancy of ≥ 12 months or > 6 months if participant has mCRPC.
* Participant is able to understand and comply with all study requirements and procedures, including completion of PRO questionnaires.
* Male participant must agree to use defined forms of contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 7 months after final ASP5541 or for 3 months after AA study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 7 months after final ASP5541 or for 3 months after AA study intervention administration.
* Male participant must not donate sperm during the treatment period and for 7 months after final ASP5541 or for 3 months after AA study intervention administration.
* Participant has adequate ventrogluteal muscle mass for an intramuscular injection.
* Participant agrees not to participate in another interventional study while receiving ASP5541 in the present study.
* Participant should have normal serum potassium (within the local laboratory normal range) at screening without supplementation.

Inclusion Criteria for Cohort 1

* Participant has been diagnosed with mCRPC documented by metastatic lesions on a bone scan, computed tomography (CT), magnetic resonance imaging (MRI) or prostate-specific membrane antigen positron emission tomography (PSMA-PET).
* Participant has evidence of disease progression defined as at least 1 of the following criteria at study entry.

  * Evidence of radiographic progression of disease prior to first dose and following the most recent prostate cancer treatment defined as PD on CT/MRI per RECIST v1.1 or on a bone scan per PCWG3.
  * PSA progression defined as an increase in PSA of at least 25% and ≥ 1 ng/mL above the nadir, confirmed by a second value at least 1 wk later, and with at least 1 of the measurements within 90 days prior to screening. PSA nadir is defined as the lowest PSA during or after the most recent treatment.
* Participant is receiving ongoing ADT with a gonadotropin-releasing hormone (GnRH) analogue or has a history of bilateral orchiectomy (i.e., surgical or medical castration). NOTE: Participants who have not had a bilateral orchiectomy must have a plan to maintain effective GnRH analogue therapy for the duration of the study.
* Participant has a serum testosterone level < 1.73 nmol/L (< 50 ng/dL) at Screening visit.
* Participant is able to swallow AA. Inclusion Criteria for Cohort 2
* Participant has been diagnosed with mHSPC documented by metastatic lesions on a bone scan, CT, MRI or PSMA-PET.
* Participant must have started castration therapy (i.e., medical or surgical) at least 14 days prior to Cycle 1 Day 1. NOTE: A participant who has not had a bilateral orchiectomy must have a plan to maintain effective GnRH analogue therapy for the duration of the study.
* Participant should have a baseline morning serum cortisol of ≥ 14 mcg/dL.
* Participant is able to swallow AA.
* For Groups B and C, participant has accessible archival tumor tissue from the primary tumor (preferred) or metastatic site (excluding bone) for which source and availability have been confirmed prior to study treatment.

Exclusion Criteria:

* Participant has any concurrent disease, infection or comorbid condition that interferes with the ability of the participant to participate in the study, which places the participant at undue risk or complicates the interpretation of data.
* Participant has known active central nervous system (CNS) metastases. NOTE: a participant with CNS metastases that have been treated with surgery and/or radiation therapy, who is no longer taking pharmacologic doses of glucocorticoids and is neurologically stable, is eligible.
* Participant has a known additional malignancy beyond prostate cancer that requires active treatment, with the exception of any of the following:

  * Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin or in situ carcinoma of any type
  * Adequately treated Stage I cancer from which participant is currently in remission and has been in remission for ≥ 2 years
  * Any other cancer from which participant has been disease-free for ≥ 5 years
* Participant has any unresolved National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) (v5.0) Grade > 2 toxicity at the Screening visit. NOTE: A participant receiving ongoing hormone replacement therapy for endocrine immune-related AEs without clinical symptoms will not be excluded.
* Participant has had major surgery (e.g., requiring general anesthesia) within 90 days before screening, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to participate in the study.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 28 days prior to Cycle 1 Day 1.
* Participant received a blood transfusion within 1 month of Cycle 1 Day 1.
* Participant has a history of impaired pituitary or adrenal gland function (e.g., Addison's disease, Cushing's syndrome).
* Participant has hemoglobin A1c (HbA1c) > 10% and was previously diagnosed with diabetes mellitus. Participant has HbA1c > 8% and was not previously diagnosed with diabetes mellitus (excluded participants may be rescreened after referral and evidence of improved control of their condition).
* Participant has jaundice or known current active liver disease from any cause, including hepatitis A (hepatitis A virus immunoglobulin M (IgM) positive, but testing for hepatitis A in screening is not required), hepatitis B [hepatitis B surface antigen (HBsAg) positive, or hepatitis B virus (HBV) DNA positive if HBsAg negative/anti-HBc positive]), or hepatitis C virus (HCV) antibody positive, confirmed by HCV RNA).
* Participant has moderate or severe hepatic impairment (Child-Pugh Class B or C).
* Participant has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by a local health authority.
* Participant has a body mass index > 40 kg/m2.
* Participant has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria within 2 yrs before screening.
* Participant has received treatment with glucocorticoids greater than the equivalent of 10 mg per day of prednisone within 4 wks prior to Cycle 1 Day 1. The use of topical, intraocular, inhalational, intranasal or intra-articular glucocorticoids is permitted.
* Participant received treatment with herbal medications within 4 wks prior to Cycle 1 Day 1 (e.g., saw palmetto). Participants must agree not to use herbal products during study participation.
* Participant is receiving current treatment with systemic ketoconazole or any other cytochrome 450 (CYP17) inhibitor. Participants who have received systemic ketoconazole or any other CYP17 inhibitor must have discontinued these agents ≥ 4 wks prior to Cycle 1 Day 1.
* Participant is receiving CYP2D6 substrates with a narrow therapeutic index (applies to Cohorts 1 & 2 only).
* Participant received prior systemic treatment with a strong inducer or inhibitor of CYP3A4 within 4 weeks of Cycle 1 Day 1. Concomitant use of strong inducers or inhibitors of CYP3A4 are not permitted on study.
* Participant requires use of biotin (i.e., vitamin B7) or supplements containing biotin higher than the daily adequate intake of 30 µg. NOTE: Participants who switch from a high dose to a dose of 30 µg/day or less prior to Cycle 1 Day 1 are eligible for study entry.
* Participant has received a live, attenuated vaccine within 30 days of planned start of study therapy. Examples of live, attenuated vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette Guérin and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live, attenuated vaccines and are not allowed.
* Participant is required to use any prohibited medication per List of Excluded Concomitant Medications.
* Participant has received any investigational therapy within 4 weeks (wks0 or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
* Participant has received ASP5541 (PRL-02) previously.
* Participant has absolute neutrophil count < 1500/μL, platelet count < 100,000/μL, hemoglobin < 9 g/dL (6.2 mmol/L ) or international normalized ratio (INR) ≥ 1.5 (unless participant is taking oral anticoagulants, in which case INR ≤ 2.0 is permitted) at Screening. NOTE: A participant may not have received any growth factors within 7 days or blood transfusions within 28 days prior to the hematology values obtained at Screening.
* Participant has serum total bilirubin (TBL) > 1.5 x upper limit of normal (ULN) (except participants with documented Gilbert's disease) or serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 x ULN at Screening.
* Participant does not have adequate renal function defined as a calculated creatinine clearance < 30 mL/min as determined by a validated algorithm for calculating creatinine clearance at Screening.
* Participant has serum albumin < 3.0 g/dL (30 g/L) at Screening.
* Participant has a known or suspected hypersensitivity to ASP5541, AA (Cohorts 1 and 2 only), prednisone or any components of the formulations used in the study.
* Participant has a gastrointestinal (GI) disorder affecting absorption. Exclusion Criteria for Cohort 1
* Prior treatment with a second-generation ARPI (e.g., AA, enzalutamide, apalutamide or darolutamide). NOTE: limited treatment with a second-generation ARPI in the neo-adjuvant, adjuvant or non-metastatic biochemically recurrent setting is permitted as long as there was no evidence of disease progression for at least 6 months following last dose.
* Treatment with any of the following for prostate cancer, during the indicated timeframe prior to enrollment:

  * Hormonal therapy (e.g., AR antagonists, 5 alpha reductase inhibitors, estrogens, cyproterone acetate) within 4 wks of Cycle 1 Day 1. Note: Treatment with bicalutamide within 6 wks prior to enrollment is not permitted. Treatment with GnRH agonists or antagonists is permitted.
  * Chemotherapy within 2 wks or 5 half-lives of Cycle 1 Day 1 (whichever is longer)
  * Biologic therapy within 4 wks of Cycle 1 Day 1
  * Immunotherapy within 4 wks of Cycle 1 Day 1
  * Radiation therapy (includes radioligands) within 4 wks of Cycle 1 Day 1
* Participant with a known BRCA mutation should be excluded unless they have previously received a PARPi or are not eligible for a PARPi, or a PARPi is not available.
* Participant has clinically significant cardiac disease, defined as any of the following:

  * Clinically significant cardiac arrhythmias including bradyarrhythmia, which are poorly controlled. Rate-controlled atrial fibrillation is permitted.
  * Congenital long QT syndrome.
  * QTcF ≥ 450 msec at Screening. If the QTc is prolonged in a participant with a pacemaker or bundle branch block, the participant may be enrolled in the study if confirmed by the medical monitor.
  * History of clinically significant cardiac disease or congestive heart failure greater than NYHA Class II or left ventricular ejection fraction measurement of < 50% at baseline. Participants must not have unstable angina (symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months.
  * Uncontrolled hypertension, defined as systolic BP > 160 mmHg or diastolic BP> 100 mmHg that has been confirmed by 2 successive measurements despite optimal medical management.
  * Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 3 months before start of study medication (except for adequately treated catheter-related venous thrombosis occurring > 1 month before Cycle 1 Day 1).

Exclusion Criteria for Cohort 2

* Prior treatment with a second-generation ARPI (e.g., AA, enzalutamide, apalutamide or darolutamide). Note: limited treatment with a second-generation ARPI in the neo-adjuvant, adjuvant or non-metastatic biochemically recurrent setting is permitted as long as there was no evidence of disease progression for at least 6 months following last dose.
* Participant has received any prior pharmacotherapy, radiation therapy or surgery for metastatic prostate cancer. The following exceptions are permitted:

  * Up to 4 months of ADT with GnRH agonists or antagonists or orchiectomy (within 4 months prior to Cycle 1 Day 1) with or without concurrent antiandrogens, with no radiographic evidence of disease progression or rising PSA levels prior to Cycle 1 Day 1.
  * Participant may have 1 course of palliative radiation or surgical therapy to treat symptoms resulting from metastatic disease if it was administered at least 4 wks prior to Cycle 1 Day 1. Radiotherapy to the prostate for participants with low volume metastatic disease is also permitted if it was administered at least 4 wks prior to Cycle 1 Day 1.
  * Up to 6 cycles of docetaxel therapy, with the last dose of docetaxel ≤ 2 months prior to Cycle 1 Day 1. A participant who has received docetaxel should have maintained a response to docetaxel of stable disease or better, by imaging and PSA, prior to Cycle 1 Day 1.
  * Up to 6 months of ADT with GnRH agonists or antagonists or orchiectomy with or without concurrent antiandrogens prior to Cycle 1 Day 1 if participant was treated with docetaxel, with no radiographic evidence of disease progression or rising PSA levels prior to Cycle 1 Day 1.
* Participant has clinically significant cardiac disease, defined as any of the following:

  * Clinically significant cardiac arrhythmias including bradyarrhythmia, which are poorly controlled. Rate-controlled atrial fibrillation is permitted.
  * Congenital long QT syndrome.
  * QTcF ≥ 450 msec at Screening. If the QTc is prolonged in a participant with a pacemaker or bundle branch block, the participant may be enrolled in the study if confirmed by the medical monitor.
  * History of clinically significant cardiac disease or congestive heart failure greater than NYHA Class II or left ventricular ejection fraction measurement of < 50% at baseline. Participants must not have symptomatic heart failure, unstable or new-onset angina or myocardial infarction within the past 12 months.
  * Uncontrolled hypertension, defined as systolic BP > 140 mmHg or diastolic BP > 90 mmHg that has been confirmed by 2 successive measurements despite optimal medical management. Participants may be receiving a maximum of 2 antihypertensives that were initiated at least 3 months prior to Cycle 1 Day 1.
* Arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks) within the last 12 months.

  * Venous thromboembolic events (deep vein thrombosis or pulmonary embolism) within the 3 months before start of study medication (except for adequately treated catheter-related venous thrombosis occurring > 1 month before Cycle 1 Day 1).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 218 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2032-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of androgen receptor pathway inhibitor (ARPI) -naïve metastatic castration-resistant prostate cancer (mCRPC) participants with Prostate Specific Antigen (PSA) decline ≥ 90% (Cohort 1) | Up to 37 months
  PSA will be recorded from blood sample.
Rate of no mineralocorticoid toxicity (Cohort 2 Group A, Safety run-in) | Up to 37 months
  No mineralocorticoid toxicity is defined as experiencing neither Grade ≥ 1 hypokalemia nor Grade ≥ 2 hypertension.
Proportion of metastatic hormone-sensitive prostate cancer (mHSPC) participants with prostate-specific antigen (PSA) ≤ 0.2 ng/mL (Cohort 2) | At 8 months
  PSA will be recorded from blood sample.
Dose-limiting toxicities (DLTs) (Cohort 3) | Up to Day 28
  A DLT is defined as any event meeting the DLT criteria occurring during the first 28 days of treatment regardless of attribution to the study drug unless it is clearly related to disease progress or intercurrent illness.
Number of participants with Adverse Events (AEs) (Cohort 3) | Up to 39 months
  AEs will be coded using MedDRA. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants With Serious Adverse Events (SAEs) (Cohort 3) | Up to 39 months
  An SAE is defined as any untoward medical occurrence that, at any dose: Results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is congenital anomaly/birth defect or other situations.
Number of participants with laboratory value abnormalities and/or AEs (Cohort 3) | Up to 37 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs (Cohort 3) | Up to 36 months
  Number of participants with potentially clinically significant ECG values.
Number of participants with vital sign abnormalities and/or AEs (Cohort 3) | Up to 37 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with physical exam abnormalities and/or AEs (Cohort 3) | Up to 36 months
  Number of participants with potentially clinically significant physical exam values.
Eastern Cooperative Oncology Group (ECOG) Performance Status (Cohort 3) | Up to 36 months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

SECONDARY OUTCOMES:
Radiographic progression-free survival (rPFS) | Up to 84 months
  Radiographic progression-free survival (rPFS) is deﬁned as the time from the date of randomization/ﬁrst dose date until the date of radiological progressive disease (PD) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and Prostate Cancer Working Group 3 (PCWG3) as determined by investigator or death from any cause.
Prostate-specific antigen (PSA) decline ≥ 50% from baseline | Up to 37 months
  Proportion of participants who had a PSA decline of ≥ 50% from baseline, confirmed by a second consecutive PSA assessment at least 3 weeks later.
PSA decline ≥ 90% (Cohorts 2 & 3 only) | Up to 37 months
  Proportion of participants who had a PSA decline of ≥ 90% from baseline, confirmed by a second consecutive PSA assessment at least 3 weeks later.
PSA undetectable rate (≤ 0.2 ng/mL) (Cohorts 1 & 3) | Up to 37 months
  Proportion of participants achieving a PSA level ≤ 0.2 ng/mL at any time post baseline.
PSA undetectable rate (≤ 0.02 ng/mL) | Up to 37 months
  Proportion of participants achieving a PSA level ≤ 0.02 ng/mL at any time post baseline.
Time to PSA progression per PCWG3 criteria | Up to 37 months
  Time from first dose date to the date of the first PSA value demonstrating a ≥ 25% increase and an absolute increase of ≤ 0.2 ng/mL above the nadir (i.e., the lowest PSA value observed post baseline or at baseline), which is confirmed by a second consecutive value at least 3 weeks later.
Objective response rate (ORR) | Up to 84 months
  Proportion of participants who achieved a confirmed Complete Response (CR) or Partial Response (PR) in their soft tissue disease using RECIST v1.1 criteria and PCWG3 for bone disease.
Duration of response (DOR) | Up to 84 months
  Time from first date of confirmed CR or confirmed PR until the date of radiological PD per RECIST v1.1 and PCWG3 as determined by investigator or death from any cause.
Best overall response (BOR) | Up to 84 months
  The best response derived from all time points' overall responses (CR, PR, stable disease or non-CR/non-PD [for participants with no measurable disease at baseline], PD, not evaluable and not determined in order).
Number of participants with Adverse Events (AEs) (Cohorts 1 & 2) | Up to 39 months
  AEs will be coded using MedDRA. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants With Serious Adverse Events (SAEs) (Cohorts 1 & 2) | Up to 39 months
  An SAE is defined as any untoward medical occurrence that, at any dose: Results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity is congenital anomaly/birth defect or other situations.
Number of participants with laboratory value abnormalities and/or AEs (Cohorts 1 & 2) | Up to 37 months
  Number of participants with potentially clinically significant laboratory values.
Urine potassium (Cohort 2) | Up to 37 months
  Potassium level will be recorded from urine sample.
Urine creatinine (Cohort 2) | Up to 37 months
  Creatinine level will be recorded from urine sample.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs (Cohorts 1 & 2) | Up to 36 months
  Number of participants with potentially clinically significant ECG values/cardiac monitoring.
Number of participants with vital sign abnormalities and/or AEs (Cohorts 1 & 2) | Up to 37 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with physical exam abnormalities and/or AEs (Cohorts 1 & 2) | Up to 36 months
  Number of participants with potentially clinically significant physical exam values.
ECOG Performance Status (Cohort 1 & 2 only) | Up to 36 months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.
Number of participants with testosterone suppression to ≤ 1 ng/dL, or achieves a ≥ 90% reduction from baseline | Up to 37 months
  Testosterone value will be recorded from blood sample.
Mean testosterone value by timepoint | Up to 37 months
  Testosterone value will be recorded from blood sample.
Time to pain progression | Up to 36 months
  Time to pain progression defined using pain scores from the Brief Pain Inventory - Short form (BPI-SF) and opiate analgesic use will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (12):
- United States (3):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- DE49004, Nürtingen, Baden-Wurttemberg, Germany
- Japan (6):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Harasanshin Hospital, Fukuoka
  - Osaka International Cancer Institute, Osaka
- PanOncology Trials, San Juan, Puerto Rico
- KR82008, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as compounds terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency